CLINICAL TRIAL: NCT05638360
Title: Evaluation of the Efficacy of Ru-Yi-Jin-Huang-Saan on Colles' Fracture ---a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Evaluation of the Curative Effect of Ru-Yi-Jin-Huang-Saan
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, LienCheng Lin, Deputy Director of Department of Traditional Chinese Medicine, Changhua Christian Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RYJHS
Record Dates: First submitted 2022-11-26; First posted 2022-12-06 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-08

CONDITIONS: Colles' Fracture
MeSH Terms: conditions — Colles' Fracture | interventions — Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ru-Yi-Jin-Huang-Saan (Experimental): Participants received Ru-Yi-Jin-Huang-Saan patch topically twice daily for 6 days.
  Interventions: Drug: Ru Yi Jin Huang Powder
- Placebo (Placebo Comparator): Participants received a starch patch topically twice daily for 6 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ru Yi Jin Huang Powder — Each patch contains 13g Ru Yi Jin Huang Powder and 10c.c. water.
  Other Names: golden patch
  Arms: Ru-Yi-Jin-Huang-Saan
Drug: Placebo — Each patch contains 13g starch and 10c.c. water.
  Other Names: starch
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Ru-Yi-Jin-Huang-Saan for the treatment of Colles' fracture.

DETAILED DESCRIPTION:
According to the definition of the World Health Organization, Taiwan officially entered the aged society in 2018. The population over the age of 65 exceeds 14% of the total population. Based on this, it is estimated that we will enter a super-aged society in 2026. Because the older the age, the higher the rate of bone loss, and the higher the risk of osteoporosis, the easier it is to fracture due to falls. The incidence of bone fracture is directly proportional to the aging population. Traditional Chinese Medicine(TCM) interventional fracture treatment has a long history and experience.

Many recent studies show that TCM is benefit to reduce risk of total hip replacement and has a positive influence on the prevention of osteoporotic fracture. In drug mechanism research, some Chinese herbal medicine has been proved to promote bone fracture healing . Although most of these researches have been confirmed in the laboratory, little information is available on true patients. In clinical we observe a lot of topical Chinese medicine been used after fracture, so the purpose of this thesis is to investigate the effective of topical Chinese herbal paste. This study may lead to build the usage of guideline after fracture.

ELIGIBILITY:
Inclusion Criteria:

1. People who are over 20 years old and have no lack of mental ability can understand the content of the experiment and are willing to participate in it.
2. Patients with Colles' fracture receive surgical fixation(ORIF).

Exclusion Criteria:

1. People are unable to cooperate with experiments and fill out questionnaires.
2. Patients have wounds on the back of their wrists.
3. Patients are allergic to traditional Chinese medicine for external applications or have used other traditional Chinese medicine for external applications.
4. Patients have cancer, stroke, and systemic diseases such as severe anemia, thyroid disease, uncontrolled diabetes, etc.
5. Pregnant woman.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Patient-Rated Wrist Evaluation(PRWE) scale at Day 6 | Baseline and Day 6
  The PRWE scale is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living.
  1. Pain subscale: contains 5 items each of which is further rated from 1-10. The maximum score in this section is 50 and minimum 0.
  2. Function subscale: contains total 10 items which are further divided into 2 sections i.e specific activities (having 6 items) and usual activities (having 4 items). The maximum score in this section is 50 and minimum 0.
  Possible scores range from 0 (best score) to 100 (worst score).
  Change = (Day 6 score - Baseline score)

SECONDARY OUTCOMES:
Change from Baseline in C-reactive protein(CRP) at Day 6 | Baseline and Day 6
  CRP is used primarily as an indicator of inflammation.The higher the value, the more severe the inflammation is.
  Change = (Day 6 score - Baseline score)
Change from Baseline with ultrasound at Day 6 | Baseline and Day 6
  ultrasound is used primarily as an indicator of swelling.The larger the value, the more swollen it is.
  Change = (Day 6 score - Baseline score)

CONTACTS AND LOCATIONS:
Overall Officials: LienCheng Lin, Master, Study Chair — Changhua Christian Hospital
Locations (1):
- Changhua Christian Hospital, Changhua, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siu WS, Shiu HT, Shum WT, Ko Chun H, Lau CBS, Hung Leung K, Leung Ping C. Chinese topical herbal medicine gives additive effect on pharmaceutical agent on fracture healing. J Tradit Chin Med. 2019 Dec;39(6):853-860. PMID 32186156
- [Background] Peng LH, Ko CH, Siu SW, Koon CM, Yue GL, Cheng WH, Lau TW, Han QB, Ng KM, Fung KP, Lau CB, Leung PC. In vitro & in vivo assessment of a herbal formula used topically for bone fracture treatment. J Ethnopharmacol. 2010 Sep 15;131(2):282-9. doi: 10.1016/j.jep.2010.06.039. Epub 2010 Jun 30. PMID 20600749
- [Background] Raittio L, Launonen AP, Hevonkorpi T, Luokkala T, Kukkonen J, Reito A, Laitinen MK, Mattila VM. Two casting methods compared in patients with Colles' fracture: A pragmatic, randomized controlled trial. PLoS One. 2020 May 29;15(5):e0232153. doi: 10.1371/journal.pone.0232153. eCollection 2020. PMID 32469881
- [Background] Wah JW, Wang MK, Ping CL. Construct validity of the Chinese version of the Patient-rated Wrist Evaluation Questionnaire (PRWE-Hong Kong Version). J Hand Ther. 2006 Jan-Mar;19(1):18-26, quiz 27. doi: 10.1197/j.jht.2005.10.003. PMID 16473730
- [Background] Neumaier M, Braun KF, Sandmann G, Siebenlist S. C-Reactive Protein in Orthopaedic Surgery. Acta Chir Orthop Traumatol Cech. 2015;82(5):327-31. PMID 26516948
- [Background] Sebastin SJ, Chung KC. An Asian perspective on the management of distal radius fractures. Hand Clin. 2012 May;28(2):151-6. doi: 10.1016/j.hcl.2012.03.007. PMID 22554658
- [Background] Yang NP, Chan CL, Yu IL, Lee CY, Chou P. Estimated prevalence of orthopaedic fractures in Taiwan--A cross-sectional study based on nationwide insurance data. Injury. 2010 Dec;41(12):1266-72. doi: 10.1016/j.injury.2010.05.025. Epub 2010 Jun 17. PMID 21288468
- [Background] Raudasoja L, Aspinen S, Vastamaki H, Ryhanen J, Hulkkonen S. Epidemiology and Treatment of Distal Radius Fractures in Finland-A Nationwide Register Study. J Clin Med. 2022 May 18;11(10):2851. doi: 10.3390/jcm11102851. PMID 35628978
- [Derived] Lin LC, Wang WH, Chang WK, Gao JL, Yang RC, Hsu PC, Lo LC. Evaluation of the Efficacy of the Traditional Chinese Medicine Formulation Ru-Yi-Jin-Huang-Saan on Colles Fracture After Surgery: Protocol for a Randomized, Double-Blind, Placebo-Controlled Trial. JMIR Res Protoc. 2025 Mar 5;14:e56849. doi: 10.2196/56849. PMID 40053806